CLINICAL TRIAL: NCT05592899
Title: Head and Neck Trauma Registry, Protocol ID: 032.MBSI.2021.D
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 032.MBSI.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-10-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Craniocerebral Trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective registry dataset of all adults who presented with cervical and/or skull base fractures or a subdural hematoma at Methodist Dallas Medical Center (MDMC) and had consults to the neurological surgery department beginning in January of 2016, and continuing until a statistically significant number of cases are obtained.

DETAILED DESCRIPTION:
This is a retrospective registry dataset of all adults who presented with cervical and/or skull base fractures or a subdural hematoma at Methodist Dallas Medical Center (MDMC) and had consults to the neurological surgery department beginning in January of 2016, and continuing until a statistically significant number of cases are obtained. Subjects will undergo no additional tests or procedures as part of this registry study. All patient data will be obtained from the patient's electronic health records of the hospital or clinic in a retrospective manner. The process for gathering the data will not influence treatment decisions. There will be no direct patient contact associated with inclusion in this registry study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Presenting to MDMC with cervical and/or skull base fractures or those with subdural hematomas

Exclusion Criteria:

* Do not meet the Study Inclusion Criteria laid out in section 4.1.
* Vulnerable populations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients 18 years of age or older
  * Presenting to MDMC with cervical and/or skull base fractures or those with subdural hematomas
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-08-23 (Estimated); Study Completion 2024-08-23 (Estimated)

PRIMARY OUTCOMES:
Collection of data for the Head and Neck Trauma Registry: Patient Demographics | Jan 2018 to Dec 2022
  To collect clinical data related to patient demographics
Collection of data for the Head and Neck Trauma Registry: traumatic diagnosis | Jan 2018 to Dec 2022
  traumatic diagnosis
Collection of data for the Head and Neck Trauma Registry: mechanism of injury, arterial injury, skeletal injury | Jan 2018 to Dec 2022
  mechanism of injury, arterial injury, skeletal injury
Collection of data for the Head and Neck Trauma Registry: radiographic modality and findings | Jan 2018 to Dec 2022
  radiographic modality and findings
Collection of data for the Head and Neck Trauma Registry: surgical management | Jan 2018 to Dec 2022
  surgical management (endovascular, open, none)
Collection of data for the Head and Neck Trauma Registry: disease course, treatment course, hospital course, treatment responses | Jan 2018 to Dec 2022
  disease course, treatment course, hospital course, treatment responses
Collection of data for the Head and Neck Trauma Registry: surgical and non-surgical outcomes | Jan 2018 to Dec 2022
  surgical and non-surgical outcomes
Collection of data for the Head and Neck Trauma Registry: reoperation rates for the same diagnosis | Jan 2018 to Dec 2022
  reoperation rates for the same diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Oh, MD, PhD, Principal Investigator — Methodist
Locations (1):
- Methodist Moody Brain and Spine Institute, Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided